CLINICAL TRIAL: NCT02865707
Title: Prevention of Ulcerative Colitis by Prebiotics: Efficacy and Protective Mechanisms
Brief Title: Ulcerative Colitis Relapse Prevention by Prebiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00041938
Record Dates: First submitted 2016-07-12; First posted 2016-08-12 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2020-03

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; prebiotics; b-fructans; inulin; oligofructose; intestinal microbiota
MeSH Terms: conditions — Colitis, Ulcerative | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic (Experimental): Prebiotic group will take 15 grams of prebiotic product Synergy-1 per day for 6 months. Synergy-1 is chicory-derived β-fructans inulin plus FOS (1:1). During the first two weeks the patient is advised to take 7.5 g of the product at breakfast only. Starting in week 3 until the end of the treatment the participant will take 7.5 g at breakfast and 7.5 g at dinner for a total of 6 months, or until you experience a flare.
  Interventions: Dietary Supplement: Synergy-1
- Placebo (Placebo Comparator): Placebo group will take 15 grams of maltodextrin per day for 6 months. Maltodextrin is a sugar adsorbed in the small bowel with no effect on the colonic intestinal microbiota. During the first two weeks the patient is advised to take 7.5 g of the product at breakfast only. Starting in week 3 until the end of the treatment the participant will take 7.5 g at breakfast and 7.5 g at dinner for a total of 6 months, or until you experience a flare.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Synergy-1 — Synergy-1 is chicory-derived β-fructans inulin plus FOS (1:1).
  Arms: Prebiotic
Dietary Supplement: Maltodextrin — Maltodextrin is carbohydrate adsorbed in the small bowel.
  Arms: Placebo

SUMMARY:
Ulcerative colitis (UC) is a relapsing chronic intestinal inflammation with no existing cure, that affects over 300 per 100.000 Canadians, the highest prevalence in the world. The standard drug therapies are expensive and potentially toxic, and mostly directed against the chronic inflammatory process. UC is the result of a dysbiosis between disease-inducing and protective intestinal bacteria in a genetically susceptible host. Non-digestible dietary carbohydrates (NDC) stimulate the growth of protective endogenous intestinal bacteria which ferment them into short-chain fatty acids (SCFA), some of the latter with natural anti-inflammatory properties, and are called prebiotics. The investigator was the first to report that oral intake of NDC, the dietary β-fructans inulin plus fructo-oligosaccharides (FOS), reduced colitis in a genetically-induced rat colitis model. Both inulin and FOS reduced colitis, each NDC modifying specific luminal microbiota. A small trial with the same mixture of NDC in patients with active UC relapsing on oral 5-aminosalicylic acid (5-ASA) showed a dose-dependent clinical response, confirming the translational potential of this NDC mixture.

The investigators propose a randomized placebo-controlled trial to assess if inulin plus FOS can also prevent such relapses in UC patients with inactive disease on stable maintenance drugs. Primary hypothesis is that inulin plus FOS is effective adjunct therapy to standard drugs for maintaining clinical remission. The second hypothesis is that the colonic microflora and its metabolic function, altered by inulin plus FOS, or not, mediate protection or relapse in UC. The longitudinal design of this maintenance prevention study and by serially collecting colon biopsies, stool, serum and urine within the same patient before a relapse (inflammation) occurs, would enable to identify unique changes in the intestinal microbiota, their metabolic functions and also assess effects on host-immune response that are associated with remission or before a relapse occurs during treatment with beta-fructans, or not.

DETAILED DESCRIPTION:
Objectives: Based on the efficacy of inulin plus FOS shown in experimental colitis as well as their ability to improve active human UC the investigators propose double-blind placebo controlled study using Synergy1, a 1:1 FOS/ inulin mixture, in patients in clinical remission of UC. The specific aims of this study are as follow:

1. To determine if β-fructans are effective in maintaining clinical remission in UC patients.
2. To examine the mechanisms of action of β-fructans on the intestinal microbiota composition and function and host immune response of these patients.

It is hypothesized that β-fructans will prolong remission in UC patients with inactive disease maintained on standard drug therapy and that the prebiotics beneficial effect is associated with enhanced colonic energy homeostasis as a result of specific stimulation of butyrate- and/ or other SCFA-producing microorganisms combined with improved host mucosal energy and inflammation regulation.

The proposed trial

Trial Design: A double blind placebo controlled clinical trial

Intervention and duration of treatment: All patients in the treatment group will receive chicory-derived β-fructans inulin plus FOS (1:1) ("Synergy1") for 6 months. Synergy1 will be administered as 7.5 gram dose twice a day as a pre-packaged powder added to meals and provided by Beneo-Orafti. This 15 gram daily prebiotic dose was found to be most effective in treating mild to moderately active UC in the investigator's previous pilot study. Patients in the placebo group will receive non-fermentable maltodextrin with a similar appearance, dosage and frequency as β-fructans. Patients that completed the 6 months treatment period will be monitored for disease related symptoms for additional 6 months.

Co-Intervention: Participants will continue at standard maintenance therapy for the duration of the trial. Participants will be asked to maintain their regular diet. This will be confirmed by having subjects complete the Food Frequency Questionnaire and assessing dietary intake at 0 and 6 months of the study, or at relapse, using online system. Compliance will be assessed by counts of study agent packages and by metabolomic analysis of participants serum and urine.

Specimen Samples: Fecal samples will be collected for fecal calprotectin (FC) and microbiota analysis at 0, 1, 3, 6 and 12 months, or at relapse. Colon biopsies will be collected between 15-20 cm from the anus for host mucosal response (4 biopsies), microbiota studies (4 biopsies) and histology (2 biopsies) at the start, and at 6 months, or at relapse. Urine and blood/serum will be collected for metabolomics analysis at 0, 1, 3 and 6 month of treatment, or at relapse. Colonic luminal washes will be collected at the start and at 6 months or at relapse during the sigmoidoscopy exam.

Sample Size: Ninety patients, 45 in each arm, will be needed to detect a difference of 30 % in the proportion of UC patients with clinical recurrence by 6 months with a power of 80% using a two-sided p=0.05 level test. An anticipated dropout rate for this trial will be 10%, based on previous maintenance trials, therefore the overall sample size for this trial will be 100 patients.

Outcomes:

Primary Outcome: The proportion of patients with relapse over 6 months. Relapse is defined as an increase of Mayo score of 3 or more with an endoscopy grade equal to or more than 2, and rectal bleeding for at least 3 days. The relapse rate in the prebiotic-treated group at 6 month will be compared to the relapse rate in the placebo group.

Secondary outcomes: 1) Time to relapse. 2) Patient compliance and tolerability. Compliance will be assessed as a ratio of packages (used) divided by the total packages dispensed over 6 months. Tolerability will be assessed by a validated questionnaire by Casellas et al on adverse effects such as bloating and flatulence, compliance by package, pill counting and metabolomic analysis at 3 and 6 months, or at relapse. 3) Intestinal inflammation (measured by fecal calprotectin) at baseline and months 1, 3 and 6, or at relapse. 4) Microscopic inflammation scores (0 and 6 months, or at relapse)

Basic science parameters: 1) Colonic biopsies for cytokine measurement, butyrate transporters and oxidation pathway and Mucin 2 (MUC2) mRNA expression analysis, histological assessment and characterization and quantification of the mucosa-associated microbiota; 2) Stool and urine for assessment of fecal calprotectin concentrations, the luminal microbiota and its metabolic products using pyrosequencing, quantitative PCR (qPCR) and gas chromatography (GC) and nuclear magnetic resonance (NMR); 3) Blood/serum for metabolomic analysis with GC and NMR; 4) colonic luminal wastes for assessing the Immunoglobulin G (IgG) associated microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ulcerative colitis (UC) with confirmed diagnosis by histology and endoscopy.
* Currently in clinical remission defined as total Mayo score of ≤ 2 and endoscopic score of 0 or 1) who have experienced at least one flare in the past 18 months.
* On stable doses of oral 5-ASA for 2 weeks and/or a stable doses of azathioprine and/or anti-tumor necrosis factor (anti-TNF) biologics for 2 months
* Colonic involvement of >15 cm from the anal verge.
* Ability to give valid informed consent
* For females of child bearing potential, a negative pregnancy test and an agreement to use appropriate birth control over the study period.

Exclusion Criteria:

* Crohn's disease, indetermined colitis or infectious colitis.
* Active UC, (total Mayo score of ≥ 3)
* Taking prednisone (or steroid equivalent) within 1 month of enrollment
* Used topical 5-ASA or steroids within 2 weeks of enrollment
* Using immunosuppressive treatments of 6-mercaptopurine or methotrexate
* Used antibiotics within 2 months
* Used anti-diarreal agents with the previous 3 days
* Pregnancy or lactation
* Significant chronic disorders such as severe cardiac disease, significant renal failure, severe pulmonary disease (need for oxygen)
* Active gastrointestinal infection
* Severe psychiatric disorder
* Not able to consent to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Prevention of relapse | 6 months
  The percentage of patients that experienced relapse during the treatment period in prebiotic group versus that in the placebo group. Percentage will be calculated using the number of patients that relapse divided to the total number of patients in the treatment group. Relapse is defined as an total Mayo score of 3 or more with an endoscopy grade equal to or more than 2, and rectal bleeding for at least 3 days.

SECONDARY OUTCOMES:
Time to relapse | 6 months
  The time the relapse occurs
Patient compliance | 3 and 6 month
  This will be assessed by package counting at 3 and 6 months or at relapse
Patient tolerability | 3 and 6 month
  The number of patients that experience adverse events related to treatment. This will be assessed by structured questionnaire at 3 and 6 months or at relapse
Changes in endoscopic disease activity inflammation | 0 and 6 month
  Endoscopic disease activity will be determined during sigmoidoscopy at baseline and 6 month or at relapse
Changes in fecal calprotectin | 0, 1, 3 and 6 month
  Mucosal inflammation will be determined by fecal calprotectin concentration at baseline and at months 1, 3 and 6 or during relapse
Changes in partial Mayo score | 0 and 6 month
  Partial Mayo score will be determined at baseline and at 6 months of treatment, or during a relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Levinus A Dieleman, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Armstrong HK, Bording-Jorgensen M, Santer DM, Zhang Z, Valcheva R, Rieger AM, Sung-Ho Kim J, Dijk SI, Mahmood R, Ogungbola O, Jovel J, Moreau F, Gorman H, Dickner R, Jerasi J, Mander IK, Lafleur D, Cheng C, Petrova A, Jeanson TL, Mason A, Sergi CM, Levine A, Chadee K, Armstrong D, Rauscher S, Bernstein CN, Carroll MW, Huynh HQ, Walter J, Madsen KL, Dieleman LA, Wine E. Unfermented beta-fructan Fibers Fuel Inflammation in Select Inflammatory Bowel Disease Patients. Gastroenterology. 2023 Feb;164(2):228-240. doi: 10.1053/j.gastro.2022.09.034. Epub 2022 Sep 29. PMID 36183751